CLINICAL TRIAL: NCT07209371
Title: Rifaximin Versus No Intervention in Patients With IgA Monoclonal Gammopathy of Undetermined Significance
Brief Title: Rifaximin Versus No Intervention for the Treatment of IgA Monoclonal Gammopathy of Undetermined Significance
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Rising Tide Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1125814; NCI-2025-06773 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0020984 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-10

CONDITIONS: IgA Monoclonal Gammopathy of Undetermined Significance
MeSH Terms: interventions — Rifaximin; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Rifaximin) (Experimental): Patients receive rifaximin orally (PO) three times daily (TID) for 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Drug: Rifaximin; Procedure: Biospecimen Collection
- Arm B (No intervention) (Other): Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection

INTERVENTIONS:
Drug: Rifaximin — Given PO
  Other Names: Xifaxan
  Arms: Arm A (Rifaximin)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection

SUMMARY:
This phase II trial compares the effect of rifaximin to no intervention for the treatment of IgA monoclonal gammopathy of undetermined significance (MGUS). Rifaximin is a type of antibiotic that is only used in cancer chemotherapy (antineoplastic antibiotic). It works by damaging the cell's DNA and may kill cancer cells or precancerous cells like those found with MGUS. Giving rifaximin may kill more precancerous cells in patients with IgA MGUS.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive rifaximin orally (PO) three times daily (TID) for 14 days in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.

ARM B: Patients undergo blood sample collection throughout the study.

After completion of study intervention, patients are followed up at 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Ability to understand and willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of potential study participants
* Clinical diagnosis of IgA monoclonal gammopathy of undetermined significance (MGUS) based on International Myeloma Working Group (IMWG)-2014 criteria (Rajkumar et al, Lancet Oncology, 2014)
* Agree to use adequate contraception

  * For women of child-bearing potential: prior to study entry and for the duration of study participation
  * For men: prior to study entry, for the duration of study participation, and one month after completion of rifaximin administration (for men)
* No antibiotic use in the preceding 2 weeks

Exclusion Criteria:

* Participants who are receiving other investigational agents
* Pregnant women
* Known hypersensitivity to rifaximin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | From the start of therapy, up to 90 days
  Defined as the proportion of patients with > 25% decline in clonal Ig at any point within 90 days after the initiation of drug or no intervention. Logistic regression will be conducted to evaluate the association between endpoint of interest and treatment (Arm A versus [vs] B).

SECONDARY OUTCOMES:
Proportion of patients experiencing > grade 2 adverse events | From the start of therapy, up to 90 days
  Logistic regression will be conducted to evaluate the association between endpoint of interest and treatment (Arm A vs B).

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Dhodapkar, MBBS, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No